CLINICAL TRIAL: NCT00243672
Title: Early Therapeutic Effects of Statins and Fibrates on Unstable Atherosclerotic Plaques: a Randomised Microarray-Study on Endarterectomy Specimens of Human Carotid Arteries
Brief Title: Early Therapeutic Effects of Statins and Fibrates on Unstable Atherosclerotic Plaques
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study chair changed his employment, the realization of the study was not possible
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-Anast-05
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin; Gemfibrozil

INTERVENTIONS:
Drug: Atorvastatin
Drug: Gemfibrozil

SUMMARY:
Rupture of unstable atherosclerotic plaques is the underlying pathophysiologic mechanism of acute coronary syndromes and thus also of perioperative myocardial ischemia. Lipid lowering drugs such as statins and fibrates have been shown to improve the outcomes of patients with atherosclerosis. This is not only mediated through their therapeutic actions on lipid metabolism, but relies on a multitude of pleiotropic effects of these substances. One of the most interesting of these effects is the stabilisation of atherosclerotic plaques.

To investigate these effects in a perioperative setting, patients scheduled for thromboendarterectomy of the carotid artery will be recruited. They will be randomised to receive either atorvastatin 10mg/d, gemfibrozil 1200mg/d or placebo for two weeks preoperatively. Specimens of carotid plaques will be obtained intraoperatively. After microscopic characterisation of plaques, DNA-microarray analyses will be done to gain insights into the transcriptional regulation and expression profiles of various types of atherosclerotic plaques under different pharmacological circumstances (stable or unstable with statin/fibrate/placebo).

ELIGIBILITY:
Inclusion Criteria:

* atherosclerosis
* stenosis of carotid artery

Exclusion Criteria:

* therapy with statine or fibrate
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Study Completion 2007-10

PRIMARY OUTCOMES:
expression profile in atherosclerotic plaque

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Theilmeier, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Münster